CLINICAL TRIAL: NCT04083222
Title: A Double-Blind, Placebo-Controlled, Phase 2 Study to Assess the Safety, Tolerability and Efficacy of IONIS-AGT-LRx, an Antisense Inhibitor Administered Subcutaneously for 8 Weeks to Hypertensive Subjects With Uncontrolled Blood Pressure
Brief Title: A Study to Assess the Safety, Tolerability and Efficacy of IONIS-AGT-LRx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 757456-CS3
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Hypertension
Keywords: Hypertension; Hypertensive; AGT; Angiotensinogen; Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received ISIS 757456-matching placebo, subcutaneous (SC) injection, once-weekly for 8 weeks and an additional loading dose on Day 3.
  Interventions: Drug: Placebo
- ISIS 757456 (Experimental): Participants received ISIS 757456 80 mg, SC injection, once-weekly for 8 weeks and an additional loading dose on Day 3.
  Interventions: Drug: ISIS 757456

INTERVENTIONS:
Drug: Placebo — ISIS 757456-matching placebo solution administered as SC injection.
  Arms: Placebo
Drug: ISIS 757456 — ISIS 757456 administered as SC injection.
  Arms: ISIS 757456

SUMMARY:
This study evaluated the effect of ISIS 757456 (IONIS-AGT-LRx) on plasma angiotensinogen (AGT) and systolic blood pressure (SBP) in uncontrolled hypertensive participants who were on two to three antihypertensive medications.

DETAILED DESCRIPTION:
This study was a Phase 2, double-blind, randomized, placebo-controlled study in 26 participants. Participants were randomized in a 2:1 ratio and received a once-weekly subcutaneous (SC) treatment with either IONIS-AGT-LRx or placebo, with an additional loading dose administered on Study Day 3. The treatment lasted for 8 weeks and the post-treatment period lasted for 13 weeks.

ELIGIBILITY:
Inclusion criteria:

* Males or females aged 18-75 inclusive and weighing ≥ 50 kilograms (kg) at the time of informed consent
* Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal
* Males must be surgically sterile or, abstinent or, if engaged in sexual relations with a woman of child-bearing potential (WOCBP), the participant or participant's non-pregnant female partner must be using a highly effective contraceptive method
* Body mass index (BMI) ≤ 35.0 kg/square meter (m^2)
* Participant must have been diagnosed with essential hypertension for a minimum of 3 months prior to screening
* At screening, the participant must have been on a stable regimen of 2 to 3 antihypertensive medications for at least 1 month prior to screening and will be required to maintain this regimen throughout the study, using either an angiotensin-converting enzyme inhibitor (ACEi) or an angiotensin II receptor blocker (ARB), as well as 1 or 2 additional antihypertensive medications in the following categories: beta blocker, acebutolol, atenolol, betaxolol, bisoprolol, carvedilol, labetalol, metoprolol, nadolol, nebivolol, propranolol, pindolol, calcium channel blocker or, non-potassium sparing diuretic

Exclusion Criteria:

* Clinically significant abnormalities in medical history, screening laboratory results, or physical examination that would render the participant unsuitable for inclusion
* History of secondary hypertension (HTN)

The use of the following at time of screening and during the course of the study:

* Other medications for the treatment of HTN (e.g., clonidine, guanfacine, guanabenz, alpha-methyldopa, hydralazine, minoxidil, diazoxide, renin inhibitors)
* Medications that may cause hyperkalemia (e.g., cyclosporine or tacrolimus, pentamidine, trimethoprim-sulfamethoxazole, all heparins)
* Oral or SC anticoagulants (e.g., warfarin, rivaroxaban, apixaban, heparin, lovenox)
* Organic nitrate preparations (e.g., nitroglycerin, isosorbide mononitrate, isosorbide dinitrate, or pentaerythritol)
* Phosphodiesterase 5 inhibitors (e.g., sildenafil, tadalafil, vardenafil, avanafil)
* Potassium-sparing diuretics (e.g., eplerenone, spironolactone, amiloride, triamterene)

Unstable/underlying cardiovascular disease defined as:

* Any history of congestive heart failure (New York Heart Association [NYHA] class II-IV)
* Any history of previous stroke, transient ischemic attack, unstable or stable angina pectoris, or myocardial infarction prior to screening
* 12-lead electrocardiogram (ECG) corrected using Fridericia's formula (QTcF) > 450 milliseconds (msec) in males and > 470 msec in females at screening, or a history or evidence of long QT syndrome
* Any clinically significant active atrial or ventricular arrhythmias
* Any history of coronary bypass or percutaneous coronary intervention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Central Alabama Research, Birmingham, Alabama
  - National Research Institute - Wilshire, Los Angeles, California
  - Orange County Research Center, Tustin, California
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Ohio Clinical Research - Lyndhurst, Lyndhurst, Ohio
  - Juno Research, LLC, Houston, Texas
  - York Clinical Research LLC, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 9 investigative sites from 13 November 2019 to 20 July 2020.
Pre-assignment Details: A total of 64 participants were screened out of which 26 were enrolled and randomized in 2:1 ratio to receive either ISIS 757456 80 mg or placebo.
Period: Overall Study
Arm/Group | Placebo | ISIS 757456
Started | 8 | 18
Completed | 8 | 16
Not Completed | 0 | 2
Not completed — Voluntary Withdrawal | 0 | 1
Not completed — Reason not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Placebo: Participants received ISIS 757456-matching placebo, SC injection, once-weekly for 8 weeks and an additional loading dose on Day 3.
- Total: Total of all reporting groups
Arm/Group | Placebo | ISIS 757456 | Total
Number analyzed (Participants) | 8 | 18 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (10) | 60 (8) | 60 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 14 | 20
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 8 | 10
  Not Hispanic or Latino | 6 | 10 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 4 | 15 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Plasma Angiotensinogen (AGT) [Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)] — Population: Per Protocol Set (PPS) included all randomized participants who had at least 1 post-baseline efficacy or exploratory measurement, received at least 7 of the 9 doses of study drug, did not alter antihypertensive medications during the treatment period and prior to Day 57, and had no significant protocol deviations that would have been expected to affect efficacy or exploratory assessments.
  micrograms per milliliter (μg/mL)
    number analyzed (Participants) | 8 | 16 | 24
    (all) | 25.5 (4.4) | 25.2 (3.4) | 25.3 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Plasma Angiotensinogen (AGT) at Day 57 Compared to Placebo
Description: The baseline for plasma AGT was defined as the average of all values prior to the first dose of study drug.
Time Frame: Baseline up to Day 57 (start of Week 9)
Population: PPS included all randomized participants who had at least 1 post-baseline efficacy or exploratory measurement, received at least 7 of the 9 doses of study drug, did not alter antihypertensive medications during the treatment period and prior to Day 57, and had no significant protocol deviations that would have been expected to affect efficacy or exploratory assessments.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | ISIS 757456
Number analyzed (Participants) | 8 | 16
percent change | -3.4 (17.8) | -67.4 (14.1)
Statistical Analysis 1: Comparison: Placebo vs ISIS 757456; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using Analysis of Variance (ANOVA) with treatment and screening angiotensin-converting enzyme inhibitor/ angiotensin receptor blockers (ACEi/ARB) dose status stratification factor

2. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Each Scheduled, Post-Baseline Visit
Time Frame: Baseline, Days 3, 8, 15, 22, 29, 36, 43, 50, 57, 64, 78, 92, 120, and 141
Population: PPS included all randomized participants who had at least 1 post-baseline efficacy or exploratory measurement, received at least 7 of the 9 doses of study drug, did not alter antihypertensive medications during the treatment period and prior to Day 57, and had no significant protocol deviations that would have been expected to affect efficacy or exploratory assessments. 'Number analyzed' indicates the number of participants with available data at the specific timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | ISIS 757456
Number analyzed (Participants) | 8 | 16
mmHg
  Baseline | 152 (8) | 153 (10)
  Change From Baseline at Day 3 | -6 (15) | -12 (14)
  Change From Baseline at Day 8 | -8 (9) | -14 (15)
  Change From Baseline at Day 15 | -0 (16) | -9 (13)
  Change From Baseline at Day 22 | -8 (15) | -8 (16)
  Change From Baseline at Day 29 | 3 (14) | -8 (16)
  Change From Baseline at Day 36 | 0 (15) | -13 (15)
  Change From Baseline at Day 43 | -2 (9) | -11 (12)
  Change From Baseline at Day 50 | -3 (12) | -17 (16)
  Change From Baseline at Day 57 | -5 (10) | -12 (16)
  Change From Baseline at Day 64: number analyzed (Participants) | 7 | 16
  Change From Baseline at Day 64 | -8 (16) | -16 (11)
  Change From Baseline at Day 78 | -8 (14) | -12 (13)
  Change From Baseline at Day 92 | -5 (13) | -15 (15)
  Change From Baseline at Day 120 | -3 (10) | -10 (14)
  Change From Baseline at Day 141 | 0 (13) | -11 (13)
Statistical Analysis 1: Comparison: Placebo vs ISIS 757456; Day 3; Test type: Superiority; p = 0.399, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 2: Comparison: Placebo vs ISIS 757456; Day 8; Test type: Superiority; p = 0.338, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 3: Comparison: Placebo vs ISIS 757456; Day 15; Test type: Superiority; p = 0.207, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 4: Comparison: Placebo vs ISIS 757456; Day 22; Test type: Superiority; p = 0.927, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 5: Comparison: Placebo vs ISIS 757456; Day 29; Test type: Superiority; p = 0.146, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 6: Comparison: Placebo vs ISIS 757456; Day 36; Test type: Superiority; p = 0.055, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 7: Comparison: Placebo vs ISIS 757456; Day 43; Test type: Superiority; p = 0.095, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 8: Comparison: Placebo vs ISIS 757456; Day 50; Test type: Superiority; p = 0.046, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 9: Comparison: Placebo vs ISIS 757456; Day 57; Test type: Superiority; p = 0.246, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 10: Comparison: Placebo vs ISIS 757456; Day 64; Test type: Superiority; p = 0.170, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 11: Comparison: Placebo vs ISIS 757456; Day 78; Test type: Superiority; p = 0.527, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 12: Comparison: Placebo vs ISIS 757456; Day 92; Test type: Superiority; p = 0.167, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 13: Comparison: Placebo vs ISIS 757456; Day 120; Test type: Superiority; p = 0.266, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 14: Comparison: Placebo vs ISIS 757456; Day 141; Test type: Superiority; p = 0.078, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor

3. Secondary Outcome: Absolute Change From Baseline in Plasma AGT at Each Scheduled, Post-Baseline Visit
Description: The baseline for plasma AGT was defined as the average of all values prior to the first dose of study drug
Time Frame: Baseline, Days 3, 8, 15, 22, 29, 36, 43, 50, 57, 64, 78, 92, 120, and 141
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Placebo | ISIS 757456
Number analyzed (Participants) | 8 | 16
ug/mL
  Baseline | 25.5 (4.4) | 25.2 (3.4)
  Change From Baseline at Day 3 | -1.7 (2.3) | -2.5 (4.2)
  Change From Baseline at Day 8 | -1.5 (3.1) | -9.6 (4.3)
  Change From Baseline at Day 15 | -1.6 (2.1) | -13.4 (5.7)
  Change From Baseline at Day 22 | -0.7 (1.6) | -15.7 (4.7)
  Change From Baseline at Day 29 | -0.8 (3.9) | -17.1 (4.0)
  Change From Baseline at Day 36 | -2.0 (2.6) | -17.2 (4.0)
  Change From Baseline at Day 43 | -2.9 (2.5) | -17.5 (3.7)
  Change From Baseline at Day 50 | -2.2 (3.2) | -17.7 (3.8)
  Change From Baseline at Day 57 | -1.1 (4.5) | -17.0 (4.1)
  Change From Baseline at Day 64: number analyzed (Participants) | 7 | 16
  Change From Baseline at Day 64 | -4.3 (3.7) | -15.9 (3.7)
  Change From Baseline at Day 78 | -3.0 (3.1) | -12.9 (3.9)
  Change From Baseline at Day 92 | -1.7 (3.9) | -9.8 (4.2)
  Change From Baseline at Day 120 | -3.1 (1.9) | -5.7 (4.0)
  Change From Baseline at Day 141 | -3.4 (4.7) | -5.8 (5.3)
Statistical Analysis 1: Comparison: Placebo vs ISIS 757456; Day 3; Test type: Superiority; p = 0.661, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 2: Comparison: Placebo vs ISIS 757456; Day 8; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 3: Comparison: Placebo vs ISIS 757456; Day 15; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 4: Comparison: Placebo vs ISIS 757456; Day 22; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 5: Comparison: Placebo vs ISIS 757456; Day 29; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 6: Comparison: Placebo vs ISIS 757456; Day 36; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 7: Comparison: Placebo vs ISIS 757456; Day 43; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 8: Comparison: Placebo vs ISIS 757456; Day 50; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 9: Comparison: Placebo vs ISIS 757456; Day 57; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 10: Comparison: Placebo vs ISIS 757456; Day 64; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 11: Comparison: Placebo vs ISIS 757456; Day 78; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 12: Comparison: Placebo vs ISIS 757456; Day 92; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 13: Comparison: Placebo vs ISIS 757456; Day 120; Test type: Superiority; p = 0.106, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 14: Comparison: Placebo vs ISIS 757456; Day 141; Test type: Superiority; p = 0.318, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor

4. Secondary Outcome: Percent Change From Baseline in Plasma AGT at Each Scheduled, Post-Baseline Visit
Description: The baseline for plasma AGT was defined as the average of all values prior to the first dose of study drug.
Time Frame: Baseline, Days 3, 8, 15, 22, 29, 36, 43, 50, 64, 78, 92, 120, and 141
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | ISIS 757456
Number analyzed (Participants) | 8 | 16
percent change
  Percent Change From Baseline at Day 3 | -6.6 (9.5) | -10.3 (16.6)
  Percent Change From Baseline at Day 8 | -4.8 (12.9) | -38.5 (16.6)
  Percent Change From Baseline at Day 15 | -6.6 (8.1) | -53.3 (22.1)
  Percent Change From Baseline at Day 22 | -2.4 (6.3) | -62.4 (17.9)
  Percent Change From Baseline at Day 29 | -2.8 (15.5) | -67.9 (13.5)
  Percent Change From Baseline at Day 36 | -8.1 (10.2) | -68.4 (13.9)
  Percent Change From Baseline at Day 43 | -10.6 (8.2) | -69.5 (11.3)
  Percent Change From Baseline at Day 50 | -7.9 (11.4) | -70.3 (11.1)
  Percent Change From Baseline at Day 64: number analyzed (Participants) | 7 | 16
  Percent Change From Baseline at Day 64 | -18.0 (15.5) | -63.5 (14.0)
  Percent Change From Baseline at Day 78 | -12.3 (12.2) | -51.1 (14.5)
  Percent Change From Baseline at Day 92 | -6.6 (14.5) | -38.9 (15.7)
  Percent Change From Baseline at Day 120 | -12.4 (7.7) | -22.1 (14.9)
  Percent Change From Baseline at Day 141 | -14.3 (17.4) | -22.3 (19.8)
Statistical Analysis 1: Comparison: Placebo vs ISIS 757456; Day 3; Test type: Superiority; p = 0.609, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 2: Comparison: Placebo vs ISIS 757456; Day 8; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 3: Comparison: Placebo vs ISIS 757456; Day 15; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 4: Comparison: Placebo vs ISIS 757456; Day 22; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 5: Comparison: Placebo vs ISIS 757456; Day 29; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 6: Comparison: Placebo vs ISIS 757456; Day 36; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 7: Comparison: Placebo vs ISIS 757456; Day 43; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 8: Comparison: Placebo vs ISIS 757456; Day 50; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 9: Comparison: Placebo vs ISIS 757456; Day 64; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 10: Comparison: Placebo vs ISIS 757456; Day 78; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 11: Comparison: Placebo vs ISIS 757456; Day 92; Test type: Superiority; p < 0.001, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 12: Comparison: Placebo vs ISIS 757456; Day 120; Test type: Superiority; p = 0.112, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor
Statistical Analysis 13: Comparison: Placebo vs ISIS 757456; Day 141; Test type: Superiority; p = 0.371, ANOVA — P-value was analyzed using ANOVA with treatment and screening ACE/ARB dose status stratification factor

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to end of post-treatment period (Day 141)
Description: Safety set included all participants who were randomized and received at least 1 dose of study drug.
Arm/Group | Placebo | ISIS 757456
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/18
Other Adverse Events (participants affected / at risk) | 3/8 | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | ISIS 757456 (N=18)
Nasopharyngitis (Infections and infestations) | 0 | 2
Urinary tract Infection (Infections and infestations) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Injection site erythema (General disorders) | 0 | 1
Injection site pruritis (General disorders) | 0 | 1
Injection site rash (General disorders) | 0 | 1
Confusion (Injury, poisoning and procedural complications) | 1 | 0
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Genitourinary symptom (Renal and urinary disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT04083222/Prot_SAP_000.pdf